CLINICAL TRIAL: NCT06671015
Title: A Prospective Randomized Controlled Trial Comparing High-Flow Nasal Cannula Versus Noninvasive Ventilation on Reintubation and Post-Extubation Respiratory Failure in High-Risk Patients With Systolic Heart Failure
Brief Title: A Trial Comparing High-Flow Nasal Cannula Versus Noninvasive Ventilation on Reintubation and Post-Extubation Respiratory Failure in High-Risk Patients With Systolic Heart Failure
Acronym: EXTUBATE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Fisher & Paykel Healthcare Limited (Unknown)
Responsible Party: Principal Investigator, Elliott Miller, Assistant Professor of Medicine, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000038572
Record Dates: First submitted 2024-10-28; First posted 2024-11-04 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-01

CONDITIONS: Systolic Heart Failure; Respiratory Failure
MeSH Terms: conditions — Heart Failure, Systolic; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients with systolic heart failure admitted to the CICU or MICU at Yale New Haven Hospital who require IMV for >24 hours.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Extubation to HFNC (Experimental): Immediately after planned extubation, the patients assigned to the HFNC group will be continuously treated by HFNC at a flow at the maximally tolerated level for 24 hours.
  Interventions: Device: Airvo 3
- Control: Extubation to NIV for 24hrs post-extubation. (Active Comparator): The NIV will be immediately initiated after planned extubation using specific, predetermined ventilator settings for 24 hours.
  Interventions: Device: Airvo 3

INTERVENTIONS:
Device: Airvo 3 — Provides effective therapy for acute hypoxemic respiratory failure and post-extubation respiratory support for 24 hours post-extubation.

SUMMARY:
This prospective, open-label randomized controlled pilot trial will enroll participants at the Yale New Haven Hospital. Patients with systolic heart failure, defined as an ejection fraction ≤40%, who require invasive mechanical ventilation (IMV) and are admitted to either the cardiac intensive care unit (CICU) or medical ICU (MICU) will be included.

Subjects meeting eligibility criteria will be randomized 1:1 to one of the two treatment groups:

* Intervention: Extubation to high-flow nasal cannula (HFNC)
* Control: Extubation to non-invasive ventilation (NIV)

DETAILED DESCRIPTION:
The primary objective is to compare the rates of reintubation and post-extubation respiratory failure for high-risk patients with systolic heart failure extubated to HFNC or NIV. Reintubation will be at the discretion of the attending physician. In doing so, this pilot study will provide the framework for an appropriately powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or non-pregnant female greater than or equal to 18 years of age
* The patient is ventilated for greater than 24 hours
* The patient has a systolic left ventricular dysfunction defined as an ejection fraction less than or equal to 40%
* The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC).

Exclusion Criteria:

* Patients actively being treated for a COPD exacerbation or known hypercapnia (PaCO2>45) on last Arterial Blood Gas (ABG)
* Patients agitated or uncooperative state
* Patients with do-not-resuscitate orders
* Patients presenting with tracheostomies or anatomical abnormalities interfering with mask fit
* Patients are prisoners
* Patient self-extubates
* Patients with pre-existing NIV prescription (e.g., obstructive sleep apnea, neuromuscular disorders, advanced COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with reintubation or respiratory failure within 72 hours post-extubation | up to 72 hours post-extubation
  Number of participants with reintubation or respiratory failure within 72 hours post-extubation

SECONDARY OUTCOMES:
Incidence of Reintubation or respiratory failure | 48 hours, 7 days, and up to ICU discharge (an average of 30 days post-extubation)
  Number of participants that experience reintubation or respiratory failure (per specific, predetermined criteria) within 48 hours, 7 days, and up to ICU discharge (an average of 30 days)
Patient intolerance to assigned treatment | up to 24 hours post-extubation
  Intolerance will be measured as the ability to continue the therapy for the 24 hour treatment period (yes/no).
Mean length of stay | up to 30 days post-extubation
  Mean length of ICU and hospital stay in days
Incidence of ICU mortality | up to ICU discharge (an average of 30 days post-extubation)
  Number of participants with mortality while in ICU
Hospital mortality | 48 hours, 72 hours, 7 days, and hospital discharge (an average of 30 days post-extubation)
  Number of participants with mortality while in hospital
Time to reintubation | Immediately post-extubation up to 30 days post-extubation
  Mean number of hours to reintubation after extubation
Respiratory rate-oxygenation (ROX) index and vector | on day of extubation
  The ROX index, defined as the ratio of oxygen saturation as measured by pulse oximetry (SpO2)/ fraction of inspired oxygen (FIO2) to respiratory rate (RR), is used as a predictor of the need to intubate in patients that received HFNC oxygen therapy. Low ROX index (< 3): Indicates a higher risk of HFNC failure. High ROX index (> 4.88): Suggests a lower risk of HFNC failure.

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Miller, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital (CICU or MICU), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No